CLINICAL TRIAL: NCT05622669
Title: Understanding Patterns of Fatigue in Health and Disease
Acronym: FATIGUE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: University of Cambridge (Other); University of Glasgow (Other); Lancaster University (Other); University of Southampton (Other); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 2-090-22
Record Dates: First submitted 2022-11-03; First posted 2022-11-18 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-02

CONDITIONS: Myeloma; Long COVID; Heart Failure
MeSH Terms: conditions — Neoplasms, Plasma Cell; Post-Acute COVID-19 Syndrome; Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Myeloma: Individuals experiencing fatigue related to myeloma or its treatment
  Interventions: Other: Observational
- Long COVID: Individuals experiencing fatigue related to Long COVID
  Interventions: Other: Observational
- Heart failure: Individuals experiencing fatigue related to heart failure or its treatment
  Interventions: Other: Observational
- Controls: Individuals who are not experiencing problematic fatigue and who do not have myeloma, long COVID, or heart failure
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Sensed and lived experience data from all groups without a specific behavioural or drug intervention

SUMMARY:
Fatigue is a common symptom and can be the most distressing symptom of a range of medical conditions. This Ecological Momentary Assessment study will investigate lived experiences of fatigue in detail in individuals with myeloma, long COVID, heart failure, and in healthy controls without fatigue.

Participants will wear ECG patches and wrist-worn sensors that measure heart rate variability, activity levels, posture, and other parameters. They will self-rate their levels of fatigue four times daily and on-demand (when fatigue levels are noticeably good or troublesome). They will participate in an end of study interview and will have an optional feedback session with a researcher to make sense of the data they have provided.

DETAILED DESCRIPTION:
Fatigue can be the most disabling symptom experienced by patients with a wide range of diseases. In primary care, it is very challenging for clinicians to differentiate between physiological fatigue (i.e., "normal" tiredness associated with lifestyle factors) and fatigue caused by underlying pathology such as heart disease or cancer. Treatment of persistent fatigue is usually by trial-and-error without attention to personalized triggers or disparate fatigue mechanisms.

This feasibility study will investigate patient experiences of fatigue in depth, combining objective measures of sensed physiological parameters with patient reports and validated patient reported outcome measures. Patients will be recruited with three distinct clinical conditions: myeloma; long COVID; and heart failure. A healthy control group will also be recruited.

Participants will participate in a feasibility study with a longitudinal, Ecological Momentary Assessment (EMA) design, wearing sensors, and providing four times daily short self-reports of fatigue over a two-to-four week period (to be determined by the individual participant and their preferences and patterns of fatigue). They will complete validated fatigue, affect, and interoceptive awareness scores at baseline and at two weeks and participate in end of study telephone interviews with a Research Assistant.

Sensors will measure objective parameters including activity levels; heart rate; sleep; and posture (sitting/standing). Additional sensors ("beacons") will measure participant's movements and positioning within their own environment (position relative to the beacons - beacon location to be determined by participant placement); environmental temperature; noise and light levels.

Data will be analysed using multilevel modelling and Machine Learning to detect patterns in the fatigue experiences and to compare fatigue measurements within individuals; between individuals with the same clinical condition; and between groups of individuals with different clinical conditions/controls.

This feasibility study will provide data that helps to determine:

* The utility and usefulness of different sensed parameters in understanding the fatigue experience
* The practicality and acceptability of collecting the proposed sensed and self-reported data and recruitment and retention rates (to inform a larger study)
* Whether there might be meaningful differences in fatigue between individuals and groups of individuals with distinct medical conditions
* Whether there is scope for a larger study into clinical "phenotypes" of fatigue (distinct classes of fatigue that might vary according to different combinations of physiological signatures, different patient descriptions/language used to describe the experience, diurnal variation, etc.)

ELIGIBILITY:
Inclusion Criteria:

* For all groups, participants will be included if they are willing to participate in intermittent ecological momentary assessments of fatigue, to wear an ECG patch, to provide questionnaire responses at baseline, and the end of the study, and to participate in an end of study interview.

Inclusion Criteria for Group A, individuals with myeloma

* A confirmed diagnosis of myeloma
* Has experienced fatigue that is perceived by the participant to be worse than "normal tiredness" and that they associate with myeloma or treatment for myeloma

Inclusion Criteria for Group B, heart failure

* A formal diagnosis of heart failure
* All stages of heart failure and all aetiologies and with no specific ejection fraction cut-off
* Has experienced fatigue that is perceived by the participant to be worse than "normal tiredness" and that they associate with their cardiac disease or its treatment

Inclusion Criteria for Group C, long COVID

* Experiencing fatigue that is perceived by the participant to be worse than "normal tiredness", with or without other physical or psychological symptoms that developed during or after an infection consistent with COVID-19
* The fatigue (plus or minus any other symptoms) has continued for greater or equal to 12 weeks, and is not explained by an alternative diagnosis

Inclusion criteria for Group D, control group

• Individuals aged 18 years or over without the disease conditions specified in Groups A to C

Exclusion Criteria:

* Exclusion Criteria Applying to all participants:

  * Difficulty communicating in English
  * Adults lacking capacity to consent
  * Under 18 years of age
  * Declines to participate
  * Under investigation for or starting treatment for an endocrine, metabolic, or thyroid condition where the participant has not been established on a stable therapeutic dose of a licensed therapy for that condition
  * A confirmed diagnosis of sleep apnoea or narcolepsy
  * HADs depression and anxiety score at baseline greater than 8 on the depression questions, which might indicate untreated or undertreated depression
  * Shift work that involves overnight working between the hours of 9pm and 9am

We will not exclude patient participants in groups A to C based on the type of prescribed medications that they are taking. Instead, this will be carefully documented.

For Group A, myeloma

* Uncontrolled hypercalcaemia
* Current or previous diagnosis of heart failure or long COVID
* An active primary cancer diagnosis other than myeloma Group B Heart Failure
* A current or previous diagnosis of myeloma or long COVID
* Active cancer Group C, long COVID
* A current or previous diagnosis of myeloma or heart failure
* Active cancer Group D, Control group
* Presence of myeloma or another active cancer, heart failure, or long COVID
* One or more chronic medical conditions which are unstable, poorly controlled, AND perceived by the individual to be causing fatigue
* Persistent or severe fatigue symptoms that are perceived by the individual to be worse than "normal tiredness"
* Taking sedating medications to manage anxiety or insomnia including but not limited to benzodiazepines or "Z" drugs, zopiclone, zolpidem, and others in this British National Formulary Class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the community and from hospital haematology and cardiology clinics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive and physical fatigue screen (zero to ten point rating) | Two to four weeks (participant defined)
  Fatigue screen based on "state" items from the validated Mental and Physical State and Trait Energy and Fatigue Scale (O'Connor P. University of Georgia; 2006). Participants will self-report their fatigue at that moment (split into physical and cognitive/mental fatigue) on a 0-10 point numerical rating scale, anchored with "I feel no fatigue" = 0 and "strongest feeling of fatigue ever" = 10. Participants will be prompted to respond via an app four times daily and can also provide on-demand ratings when their fatigue levels are particularly problematic or when they are not experiencing problematic fatigue. Multilevel modelling will be conducted to identify changes in fatigue over time and to explore the relationships between self-reported fatigue scores and sleep, activity levels (step-count, posture, measured by wrist worn sensor), respiratory rate (measured by ECG patch), and heart rate variability (measured by ECG patch)
Lived experiences of fatigue interview | 1 day (End of study interview)
  Qualitative data collected by an end of study interview according to a topic schedule
Views and opinions about the sensing technologies interview | 1 day (End of study interview)
  Qualitative data collected by an end of study interview according to a topic schedule
Views and opinions about the trial methods and study participation interview | 1 day (End of study interview)
  Qualitative data collected by an end of study interview according to a topic schedule

SECONDARY OUTCOMES:
Drop-out rate | Participant-led study end date - two to four weeks
  The proportion of participants who drop out of the study before the end of study interview

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
This project has put in place a data sharing plan in accordance with the International Committee of Medical Journal Editors (ICMJE), as published in Annals.org on 6 June 2017.
  Data will be shared with investigators whose proposed use of the data has been approved by the Research Ethics Committee and who are parties to the project data sharing agreement for the purposes of conducting analyses to achieve the aims in the approved protocol. The data will be made available as pseudonymised data shared using a University of Aberdeen approved data sharing platform.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data sharing will start in December 2022 and data sharing may continue until the end of the retention period for research data generated by the study (current retention period 20 years).
Access Criteria: Party to the project data sharing agreement Use approved by Research Ethics Committee.

REFERENCES:
- [Derived] Adam R, Lotankar Y, Sas C, Powell D, Martinez V, Green S, Cooper J, Bradbury K, Sive J, Hill DL. Understanding patterns of fatigue in health and disease: protocol for an ecological momentary assessment study using digital technologies. BMJ Open. 2024 May 27;14(5):e081416. doi: 10.1136/bmjopen-2023-081416. PMID 38802273

DOCUMENTS (1):
  • Informed Consent Form (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT05622669/ICF_000.pdf